CLINICAL TRIAL: NCT00331929
Title: Respiratory Health Study of Children in Kiryat Tivon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Haim Bibi, Carmel Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Ped-2/2006; HTA 3653; CMC 06013904
Record Dates: First submitted 2006-05-28; First posted 2006-05-31 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2007-12

CONDITIONS: Bronchial Asthma; Signs and Symptoms, Respiratory; Allergy
Keywords: Asthma; Allergy; Respiratory; Pollution; Children; Air pollution
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Cohort of school children that evaluated with questionnaire and spirometry with MINATO 500 JAPAN spirometer
  Interventions: Device: Minato A 500 AS spirometer

INTERVENTIONS:
Device: Minato A 500 AS spirometer — Spirometry at rest
  Other Names: Spirometer MINATOm AS 500 JAPAn

SUMMARY:
Kiryat Tivon is located close to a major industrial zone. The aim of the study is to evaluate the health status of children living in K. Tivon.

The health status will be evaluated using health questionnaires and spirometry.

DETAILED DESCRIPTION:
Kiryat Tivon is located close to a major industrial zone. The aim of the study is to evaluate the health status of children living in K. Tivon.

The health status will be evaluated while using health questionnaires and spirometry.

Objective: To evaluate the respiratory health of K. Tivon children with comparatives, with respect to local air pollution levels.

Material and Methods: All the school children from K. Tivon (1800 children) will be included in the study, after both parents and the children (above 12 years of age) will sign an informed consent form.

First step: A health questionnaire (based on Hebrew version of ISAAC questionnaire) will be filled in by the parents.

Second step: Spirometry checking of the children.

In parallel, air pollution levels will be measured and provided by a network of ground monitoring stations maintained by the Haifa District Municipality Association for the Environment (HDMAE). The station provides half-hourly measurement of mean concentrations of gaseous (NOX, SO2, O3) and particular (PM 10) pollutants over the entire investigation window. Additional meteorological data are also collected.

Risk maps: Using a GIS platform, we are developing a multi-layer risk mapping procedure which accounts for ambient concentrations of selected pollutants and the heterogenic spatial distribution of several demographic and socio-economic indexes in the region.

The prevalence of pulmonary disease will be evaluated according to the risk maps.

ELIGIBILITY:
Inclusion Criteria:

* All school children

Exclusion Criteria:

* Children that their parents did not signed the informed consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 638 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The prevalence of respiratory symptoms in respect to air pollution | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Haim Bibi, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Elementary School, Kiryat Tiv'on, Israel

REFERENCES:
- [Background] Schwartz J. Air pollution and children's health. Pediatrics. 2004 Apr;113(4 Suppl):1037-43. PMID 15060197
- See also: air pollution and asthma — http://www.arb.ca.gov/research/asthma/asthma.htm